CLINICAL TRIAL: NCT07064408
Title: Effects of Subanesthetic Dose of Esketamine on Hemodynamic Stability and Postoperative Recovery Quality in Elderly Thoracic Surgery Patients Under General Anesthesia: A Randomized Controlled Clinical Trial
Brief Title: Subanesthetic Esketamine for Hemodynamic Stability and Recovery in Elderly Thoracic Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023026
Record Dates: First submitted 2025-06-25; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Hemodynamic Instability; Postoperative Recovery; Thoracic Surgery; Anesthesia, General; Elderly Patients
Keywords: Esketamine; Hemodynamic stability; Anesthesia induction; Recovery quality; Elderly patients; Thoracic surgery; Postoperative outcomes; Randomized controlled trial; Perioperative management
MeSH Terms: interventions — Esketamine; Saline Solution; Sodium Chloride; Midazolam; Sufentanil; Propofol; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine Group (Experimental): Participants in this group received a subanesthetic dose of esketamine (0.25 mg/kg) intravenously during induction of general anesthesia. The esketamine was administered slowly over approximately 30 seconds after midazolam and sufentanil, and prior to propofol and rocuronium. Standard anesthesia induction and maintenance protocols were followed thereafter.
  Interventions: Drug: Esketamine; Drug: Midazolam; Drug: Sufentanil; Drug: propofol; Drug: Rocuronium
- Control Group (Placebo Comparator): Participants in this group received an equivalent volume of 0.9% normal saline intravenously during induction of general anesthesia, administered in the same manner and time frame as in the esketamine group. The saline was administered after midazolam and sufentanil, and prior to propofol and rocuronium. All other aspects of anesthesia management were identical to the esketamine group.
  Interventions: Drug: Normal Saline (0.9% Sodium Chloride); Drug: Midazolam; Drug: Sufentanil; Drug: propofol; Drug: Rocuronium

INTERVENTIONS:
Drug: Esketamine — Intravenous administration of a subanesthetic dose of esketamine (0.25 mg/kg) during induction of general anesthesia. The drug was administered slowly over approximately 30 seconds after midazolam (2 mg) and sufentanil (50 µg), and prior to propofol (2 mg/kg) and rocuronium (0.6 mg/kg). The goal was to evaluate its effect on intraoperative hemodynamic stability and postoperative recovery in elderly patients undergoing thoracic surgery.
  Arms: Esketamine Group
Drug: Normal Saline (0.9% Sodium Chloride) — Intravenous administration of an equivalent volume of 0.9% normal saline during anesthesia induction, matching the timing and method of the esketamine group. Used as a placebo comparator.
  Arms: Control Group
Drug: Midazolam — Intravenous administration of 2 mg midazolam during anesthesia induction for sedation. Administered prior to study drug.
Drug: Sufentanil — Intravenous administration of 50 µg sufentanil for analgesia during anesthesia induction. Administered prior to study drug.
Drug: propofol — Intravenous administration of 2 mg/kg propofol for loss of consciousness during anesthesia induction. Administered after study drug.
Drug: Rocuronium — Intravenous administration of 0.6 mg/kg rocuronium to facilitate neuromuscular blockade and endotracheal intubation.

SUMMARY:
This retrospective study evaluated the effects of a subanesthetic dose of esketamine (0.25 mg/kg) on intraoperative hemodynamic stability and postoperative recovery quality in elderly patients (aged 65-75) undergoing thoracic surgery under general anesthesia. A total of 230 patients were included and randomly assigned to receive either esketamine or placebo during anesthesia induction. Key outcomes included blood pressure and heart rate stability, catecholamine levels, recovery time, incidence of adverse events such as delirium or nausea, and opioid use.

DETAILED DESCRIPTION:
Elderly patients are at increased risk for anesthesia-related complications due to reduced physiological reserves and comorbidities. Thoracic surgery further increases this risk by inducing significant cardiovascular and sympathetic stress. Esketamine, the S-enantiomer of ketamine, possesses sympathomimetic and analgesic properties that may help stabilize circulation and reduce postoperative complications when used at subanesthetic doses.

In this single-center, randomized controlled trial, patients aged 65-75 scheduled for elective thoracic surgery were administered either 0.25 mg/kg esketamine or normal saline during anesthesia induction. Hemodynamic parameters (mean arterial pressure, heart rate), plasma catecholamine concentrations (norepinephrine, epinephrine), and adverse cardiovascular responses were recorded. Postoperative outcomes included emergence time, PACU stay, incidence of delirium, hallucinations, nausea and vomiting, and opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-75 years
* Scheduled for elective thoracic surgery (e.g., lobectomy, bullectomy)
* ASA physical status I-III
* Adequate cardiopulmonary function
* Able to provide informed consent
* Preoperative systolic blood pressure <160 mmHg with stable control
* No cognitive impairment

Exclusion Criteria:

* Severe cardiovascular disease (e.g., unstable angina, heart failure ≥ NYHA class III)
* History of cerebrovascular disease
* Uncontrolled hypertension (SBP >180 mmHg)
* Severe hepatic or renal dysfunction
* Chronic psychiatric illness or long-term CNS-active drug use
* Allergy to ketamine or its derivatives
* Elevated intracranial or intraocular pressure
* Use of monoamine oxidase inhibitors within 24 hours before surgery
* History of substance abuse

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum Decrease in Mean Arterial Pressure (MAP) During Anesthesia Induction | From anesthesia induction to skin incision (approximately 15 minutes)
  The lowest value of MAP recorded between the time of anesthesia induction and skin incision, compared to baseline MAP before induction. This outcome evaluates the degree of hemodynamic depression associated with induction agents and the protective effect of esketamine.

SECONDARY OUTCOMES:
Time to Eye Opening After Surgery | Postoperative period in PACU (within 30 minutes after surgery)
  The duration between the end of surgery and the patient's spontaneous eye opening, measured in minutes in the PACU.
Incidence of Hypotension During Anesthesia Induction | From anesthesia induction to intubation (approximately 5 minutes)
  Defined as mean arterial pressure (MAP) < 65 mmHg or the need for vasopressor intervention (norepinephrine) between induction and intubation.
Incidence of Postoperative Delirium | From PACU admission to hospital discharge (up to 24 hours postoperatively)
  Evaluated using the Confusion Assessment Method for the ICU (CAM-ICU) during the recovery period.
Postoperative Morphine Requirement | Within 1 hour after surgery in PACU
  Number of patients requiring morphine for pain relief and total dose (mg) administered in the PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical and privacy considerations and the absence of participant consent for data sharing.